CLINICAL TRIAL: NCT06403956
Title: The Effect of Hand Hygiene Training Given With Different Methods on Students' Hand Hygiene Beliefs, Practices and Skills
Brief Title: Students' Hand Hygiene Beliefs, Practices and Skills
Acronym: SHHBPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Banu CİHAN ERDOĞAN, RN, PhD, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BCE
Record Dates: First submitted 2024-04-25; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Complications of Medical and Surgical Care (Y62-Y84)
Keywords: Education; Hand hygiene; Home care services; Skills
MeSH Terms: interventions — Videotape Recording; Paint

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- video group (Experimental): The population of the study consisted of 123 students who were first-year students in the Home Patient Care Program. Video group (n=29)
  Interventions: Other: Training with video
- Paint group (Experimental): The population of the study consisted of 123 students who were first-year students in the Home Patient Care Program. Paint group (n=29)
  Interventions: Other: Training with paint
- Control group (No Intervention): The population of the study consisted of 123 students who were first-year students in the Home Patient Care Program. Control group (n=29)

INTERVENTIONS:
Other: Training with video — The hand washing skills of the students in the three groups were evaluated by a researcher by observing the hand washing of the students in the sink with the Hand Washing Skills Checklist. After the students were given theoretical information about hand hygiene, including the importance of hand washing, the situations in which hands should be washed, and the steps of hand washing skills, the laboratory practice was started immediately afterwards. In the laboratory, hand washing training was given to the video group with the hand washing video developed by the researchers within the scope of the course. Afterwards, the same researcher who made the first observation re-evaluated the handwashing skills of all students in the sink by filling out the Handwashing Skill Checklist.
  Arms: video group
Other: Training with paint — The hand washing skills of the students in the three groups were evaluated by a researcher by observing the hand washing of the students in the sink with the Hand Washing Skills Checklist. After the students were given theoretical information about hand hygiene, including the importance of hand washing, the situations in which hands should be washed, and the steps of hand washing skills, the laboratory practice was started immediately afterwards. In the laboratory, hand washing training was given to the paint group with the demonstration method using acrylic paint instead of soap. Afterwards, the same researcher who made the first observation re-evaluated the handwashing skills of all students in the sink by filling out the Handwashing Skill Checklist.
  Arms: Paint group

SUMMARY:
ABSTRACT This study was conducted to determine the effect of hand hygiene training given to home patient care students with different methods on their hand hygiene beliefs, practices and skills. This study was a randomized controlled trial. The population of the study consisted of 123 students. After the removals, the study was completed with 75 students in the video, paint and control groups. In the intervention of the study, lecture, discussion, question and answer, demonstration, coloring and video methods were used.

DETAILED DESCRIPTION:
Hand hygiene is the most important strategy to prevent the transmission of microorganisms between patients, healthcare personnel and the healthcare environment. This study was conducted to determine the effect of hand hygiene training given to home patient care students with different methods on their hand hygiene beliefs, practices and skills. This study was a randomized controlled trial. The population of the study consisted of 123 students. After the removals, the study was completed with 75 students in the video (n=25), paint (n=25) and control (n=25) groups. In the intervention of the study, lecture, discussion, question and answer, demonstration, coloring and video methods were used.

ELIGIBILITY:
Inclusion Criteria:

* No previous training in a health field,
* First time students taking the Care Principles and Practices Lecture
* Students who agreed to participate in the study

Exclusion Criteria:

* Previous education in one of the health fields,
* Repeatedly taking the Care Principles and Practices Lecture
* Students who refused to participate in the study

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
The Descriptive Characteristics and Hand Hygiene Information Form | 1 year
  It was developed by the researchers and includes seven questions including age, gender, family type, economic status, previous hand hygiene training, need for hand hygiene training, and hand washing frequency.
Hand Washing Skills Checklist | 1 year
  The checklist prepared by the researchers in line with the WHO (World Health Organization) guidelines consists of 20 steps to evaluate the hand washing skills of the students. For the developed checklist, expert opinion was obtained from 5 Fundamentals of Nursing experts. Among the steps in the checklist, 0 points were given to the steps that were not applied, 0.5 points to the missing applied steps, and 1 point to the correctly applied steps. The highest score that students can get from the hand washing skill checklist is 20 points.
Hand Hygiene Belief Scale and Hand Hygiene Practice Inventory | 1 year
  It was developed by Thea F. Van De Mortel (2009). The Turkish validity and reliability of the Hand Hygiene Belief Scale and Hand Hygiene Practice Inventory were conducted by Karadağ et al. The Hand Hygiene Belief Scale and Hand Hygiene Practice Inventory were used to evaluate students' hand hygiene beliefs and practices. The Hand Hygiene Belief Scale is scored as "1=strongly disagree, 2=disagree, 3=not sure, 4=agree, 5=strongly agree" and consists of 22 items in total; the Hand Hygiene Practice Inventory is scored as "1=never, 2=sometimes, 3=often, 4=most of the time, 5=always" and consists of 14 items. Items 5,8,16,17,18,19,20 are evaluated in reverse (5=strongly disagree, 4=disagree, 3=not sure, 2=agree, 1=strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Banu CIHAN ERDOGAN, PhD, Principal Investigator — Çankırı Karatekin University
Locations (1):
- Çankırı Karatekin University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Graveto JMGDN, Rebola RIF, Fernandes EA, Costa PJDS. Hand hygiene: nurses' adherence after training. Rev Bras Enferm. 2018 May;71(3):1189-1193. doi: 10.1590/0034-7167-2017-0239. English, Portuguese. PMID 29924172
- [Result] Novak M, Breznicky J, Kompanikova J, Malinovska N, Hudeckova H. Impact of hand hygiene knowledge on the hand hygiene compliance. Med Glas (Zenica). 2020 Feb 1;17(1):194-199. doi: 10.17392/1051-20. PMID 31556581
- [Result] Ojanpera H, Kanste OI, Syrjala H. Hand-hygiene compliance by hospital staff and incidence of health-care-associated infections, Finland. Bull World Health Organ. 2020 Jul 1;98(7):475-483. doi: 10.2471/BLT.19.247494. Epub 2020 May 26. PMID 32742033
- [Result] Spruce L. Hand Hygiene. AORN J. 2021 Mar;113(3):286-294. doi: 10.1002/aorn.13340. No abstract available. PMID 33646589
- [Result] Hammerschmidt J, Manser T. Nurses' knowledge, behaviour and compliance concerning hand hygiene in nursing homes: a cross-sectional mixed-methods study. BMC Health Serv Res. 2019 Aug 5;19(1):547. doi: 10.1186/s12913-019-4347-z. PMID 31382968